CLINICAL TRIAL: NCT03947125
Title: New Application of Buprenorphine Patch on Painful Knee Joint in Knee Osteoarthritis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Bum Choi, Assistant Professor, Ajou University School of Medicine
Other Study IDs: AJIRB-MED-MDB-19-069
Record Dates: First submitted 2019-05-08; First posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- knee applied group: the patients with buprenorphine patch applied to painful knee joint in knee osteoarthritic patients
  Interventions: Drug: Buprenorphine transdermal patch on knee joint
- chest applied group: the patients with buprenorphine patch applied to anterior chest wall in knee osteoarthritic patients
  Interventions: Drug: Buprenorphine transdermal patch on knee joint

INTERVENTIONS:
Drug: Buprenorphine transdermal patch on knee joint — Conventionally buprenorphine transdermal patch had been applied to anterior chest wall or upper arm. But author had applied buprenorphine transdermal patch to painful knee joint in knee osteoarthritic patients. This research is about the effect, adverse effects, and compliance of comparison conventional chest applied buprenorphine transdermal patch group with painful knee joint applied group in knee osteoarthritic patients.
  Other Names: Buprenorphine transdermal patch on chest wall

SUMMARY:
Osteoarthritis (OA) is already one of the most disabling diseases in developed countries. Intra-articular (IA) injection of opioid in joints has been widely studied for its simplicity, safety and efficacy. We suggest the method of opioid patch regional application to OA patients instead of intra-articular opioid injections. We had applied buprenorphine patch to painful knee joint in knee OA patients, and compared knee application with conventional chest application for analgesic effects, adverse effects and compliance of buprenorphine patch. We willl retrospectively enroll about 200 patients with knee OA who did not respond to conventional therapy. Numeric rating scale (NRS), adverse effects, and compliance were checked and recorded before and after buprenorphine patch applied. All parameters were compared between chest applied group and knee applied group.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is one of the most disabling diseases in developed countries. Pain is the most uncomfortable symptom, often difficult to manage because it is aggravated by weight bearing and movement of hip and knee joints. Paracetamol, traditional nonsteroidal-anti-inflammatory drugs (NSAIDs), and cyclooxygenase (COX) -2 specific inhibitors may relieve pain of joints origin. NSAIDs and COX-2 inhibitors have many potentially serious side effects, especially in elderly patients. The 2008 and 2009 guidelines now recommend weak opioids or low doses of strong opioids when paracetamol, with or without topical NSAIDs, does not relieve pain sufficiently. However, whereas several randomized controlled studies have showed analgesic effects in musculoskeletal disease, adverse effects are common, and about 50% discontinue opioid treatment because of adverse effects.

Meanwhile, intra-articular (IA) opioid injection has been studied for some time. Opioid binding receptors have been identified within synovium of joint space, suggesting that analgesic effect of opioid injected into IA space may be locally mediated. When injected at the end of arthroscopic surgery, IA opioid could reduce postoperative pain through peripheral opioid receptors. It has also been reported to reduce pain through other pathways such as inflammatory reaction.

We suggest the method of application of buprenorphine transdermal patch instead of intra-articular injection and the hypothesis that application of opioid transdermal patch on painful joint would transport opioid component to joint space by diffusion. This hypothesis had been named Jong's hypothesis after Jong Bum Choi, the originator. We had applied buprenorphine transdermal patch at painful knee joint in knee OA patients, and they had showed good analgesic effect and low adverse effects. The purpose of this research is to show the analgesic effects, adverse effects and compliance of buprenorphine transdermal patch applied on painful knee joint in knee OA patients and compare knee applied group with conventional chest applied group in all parameters.

In medical records, we will retrospectively enroll about 200 patients with OA who were not responds to conventional therapy. Inclusion criteria were as next. 1) Age over 20, 2) diagnosis of osteoarthritis of the knee by radiographic evidence of osteoarthritis of the knee, as defined by Grades II to IV of the Kellgren and Lawrence scale, 3) Pain score over 4 in NRS from the relevant joint 4) buprenorphine transdermal patch prescribed in unilateral OA of knee. Exclusion criteria were as next. 1) total knee replacement surgery history, 2) patients treated with weak or strong opioid analgesics, 3) patients had contraindications to treatment with opioid medication, such as history of alcohol or substance abuse, 4) patients had clinically significant systemic disease or any reduced organ function, 5) patient was using antidepressants, antiepileptic drug, steroids, hypnotics (that may increase respiratory depression of buprenorphine). Patients were divided two groups. One group is the patients with chest applied buprenorphine transdermal patch, and the other group is the patients with painful knee joint applied buprenorphine transdermal patch.

NRS will be checked before and next visit (at 2 weeks or 1month after prescription of buprenorphine transdermal patch). Adverse effects of buprenorphine transdermal patches will be checked and recorded. Compliance of buprenorphine transdermal patch was investigated. All parameters will be compared in chest applied group with knee applied group.

The t-test will be used to compare the chest applied group and knee applied group in demographic data. The Mann-Whitney test, Chi-squared test, and Fisher's exact test will be used to compare two groups in NRS, adverse effects, compliance and dose of buprenorphine. All statistical analyses will be performed by use of R software, version 3.5.1. A p-value less than 0.05 will be considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 20
2. diagnosis of osteoarthritis of the knee by radiographic evidence of osteoarthritis of the knee, as defined by Grades II to IV of the Kellgren and Lawrence scale
3. Pain score over 4 in NRS from the relevant joint
4. buprenorphine prescribed in unilateral OA of knee

Exclusion Criteria:

1. total knee replacement surgery history
2. patients treated with weak or strong opioid analgesics
3. patients had contraindications to treatment with opioid medication, such as history of alcohol or substance abuse
4. patients had clinically significant systemic disease or any reduced organ function
5. patient was using antidepressants, antiepileptic drug, steroids, hypnotics (that may increase respiratory depression of buprenorphine).

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We will retrospectively enroll about 200 patients with osteoarthritis who are not responds to conventional therapy
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-05-15 (Estimated); Primary Completion 2019-06-15 (Estimated); Study Completion 2019-07-30 (Estimated)

PRIMARY OUTCOMES:
Numeric rating scale after buprenorphine transdermal patch | up to 1 month
  Numeric rating scale score is from 0 to 10 point for pain measuring scale

SECONDARY OUTCOMES:
adverse effects | up to 1 month
  side effects of buprenorphine transdermal patch
compliance of buprenorphine transdermal patch | up to 1 month
  compliance is the rate of continuing the drug

IPD SHARING:
Plan to Share IPD: No